CLINICAL TRIAL: NCT06032624
Title: Comparative Study Between Ketamine and Dexmedetomidine as Additives to Local Anesthetic in Ultrasound-guided Combined Sciatic and Femoral Nerve Block
Brief Title: Ketamine and Dexmedetomidine Comparative Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Mohammed Ahmed Mahmoud, Lecturer, Sohag University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: Soh-Med-22-07-34
Record Dates: First submitted 2022-11-09; First posted 2023-09-13 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Post Operative Pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ketamine group (group K) (Active Comparator): Ketamine group (group K):40 ml 0.5%bupivacaine and 0.5 mg\kg ketamine.
  Interventions: Procedure: combined ultra-sound guided femoral and sciatic nerve block.
- Dexmedetomidine group (group D) (Active Comparator): Dexmedetomidine group (group D) 40 ml 0.5% bupivacaine and 50µg\kg dexmedetomidine.
  Interventions: Procedure: combined ultra-sound guided femoral and sciatic nerve block.

INTERVENTIONS:
Procedure: combined ultra-sound guided femoral and sciatic nerve block. — Femoral nerve block, The femoral area will be scanned behind the midpoint of the inguinal ligament and the depth of the image will be set at 3-5 cm, and a linear high frequency 8-12MHz) probe will be placed perpendicular to the course of the femoral nerve., the volume of 15 ml of bupivacaine will be injected to perform the block. Sciatic nerve block, A curvilinear low-frequency (3-9 MHz) probe will be used to do a scan of the sub-gluteal region below a line from the ischial tuberosity and greater trochanter which are seen as two hyperechoic bony prominences,A volume of 25 ml of bupivacaine will be injected to perform the block.

SUMMARY:
In this study, the investigators will compare the effect of adding ketamine and dexmedetomidine to bupivacaine in US-guided combined sciatic and femoral nerve blocks as regards the onset and duration of the block, postoperative visual analogue scale, and analgesic consumption.50 patients with American Society of Anesthesiologists (ASA) grade I to II, 18 to 60 years of age scheduled for below-knee surgeries, Will be included in the study.

DETAILED DESCRIPTION:
The patients will be randomly classified into two groups:

Ketamine group (group K):40 ml 0.5%bupivacaine and 0.5 mg\kg ketamine, Dexmedetomidine group (group D) 40 ml 0.5% bupivacaine and 50µg\kg dexmedetomidine.

Femoral nerve block: The femoral area will be sterilized using povidone-iodine and alcohol and then drapes will be put on the patient's thigh, with the operator on the right-hand side for blocks on both sides and vice versa for a left-handed operator. The ultrasound machine will be placed on the opposite side so that the operator's line of sight, the needle, and the screen are in a straight line. The femoral area will be scanned behind the midpoint of the inguinal ligament and the depth of the image will be set at 3-5 cm and a linear high frequency 8-12MHz) probe will be placed perpendicular to the course of the femoral nerve., medial to the lateral sliding movements of the transducer-aided visualization of the pulsatile femoral artery. Structures that will be visualized: fascia iliac, femoral artery, immediately below, and lateral is the femoral nerve in a wedge-shaped space. The femoral nerve typically is hyperechoic and lies in a sulcus in the iliopsoas inferiorly. In-line insertion of the needle to reach below fascia iliaca and then a volume of 15 ml of bupivacaine will be injected to perform the block.

Sciatic nerve block: The patient will be positioned with the side for the block uppermost, flexed partially at the hip and knee joints. The iliac area will be sterilized using povidone-iodine and alcohol, and then drapes will be put on the patient's thigh, with the operator on the right-hand side for blocks on both sides and vice versa for a lefthanded operator. The ultrasound machine will be placed on the opposite side so that the operator's line of sight, the needle, and the screen is in a straight line. A curvilinear low-frequency (3-9 MHz) probe will be used to do a scan of the sub-gluteal region below a line from the ischial tuberosity and greater trochanter which are seen as two hyperechoic bony prominences; the gluteus maximus muscle is as the most superficial muscular layer bridging the two osseous structures; sciatic nerve lies deep into the gluteus maximus muscle and superficial to the quadratus femoris muscle as an oval or roughly triangular hyperechoic structure. A volume of 25 ml of bupivacaine will be injected to perform the block.

The onset and duration of sensory loss and motor blockade will be studied. The loss of pinprick sensation will be checked every 5 minutes till the onset of loss of sensation and then every 2 hours till the regain of sensation. The motor blockade will be assessed every 5 minutes till the loss of movements and then every 2 hours till the regain of movements.

The onset of action: Sensory and motor blockade Sensory block: The time interval between full deposition of local anesthetic solution till loss of pinprick sensation at the site of surgery.

Motor block: The time interval between administering the local anesthetic solution to the loss of movements.

Duration of blockade:

Sensory block: Time interval between loss of pinprick sensation to the appearance of pinprick sensation.

Motor block: Time interval between loss of movements to the appearance of the movements.

The basal heart rate (HR); noninvasive arterial systolic blood pressure (SBP) and diastolic blood pressure (DBP); and peripheral oxygen saturation (SpO2) will be recorded. An 18-gauge (G) i.v. the cannula will be inserted in the non-operated arm and lactated Ringer's solution will be started at 5 ml/kg/h.

HR, SBP, and DBP will also be recorded at 0, 5, 10, 15, 30, 45-, 60-, 90-, and 120-min. Adverse effects will be considered as hypotension (i.e., 20% decrease relative to baseline), bradycardia (HR <50 beats/min), nausea, vomiting, and hypoxemia (SpO2 <90%). Any need for additional medication will be noted intraoperatively. Blood loss will be calculated by the gravimetric method and will be replaced if more than the allowable blood loss. Pain will be assessed using a visual analog scale (VRS) (O=no pain 1=mild pain 2=moderate pain 3=severe pain 4=unbearable pain).

ELIGIBILITY:
Inclusion Criteria:

50 patients with American Society of Anesthesiologists (ASA) grade I to II, 18 to 60 years of age scheduled for below-knee surgeries, Will be included in the study.

-

Exclusion Criteria:

* Patient refusal.
* Patient with significant neurological, psychiatric or neuromuscular disease.
* Alcoholism.
* Drug abuse.
* Pregnancy or lactating women.
* Suspected Coagulopathy.
* Morbid obesity.
* Known allergy to study medications.
* Septicaemia and local infection at the block site.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-12-01 (Estimated); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
the onset of the femoral nerve block | from the deposition of the local anesthetic till the loss of pinprick sensation
  The time interval between the deposition of the local anesthetic and the loss of pinprick sensation at the site of surgery.